CLINICAL TRIAL: NCT05040269
Title: Serum Levels of Vitamine D,Calcium and Magnesium in Infants and Preschool Children With Recurrent Wheezing
Brief Title: Serum Levels of Vitamin D,Calcium and Magnesium in Preschool Recurrent Wheezers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Samar Alsoudy Ahmed, Resident doctor at pediatric department sohag university hospital, Sohag University
Other Study IDs: Soh-Med-21-07-04
Record Dates: First submitted 2021-08-22; First posted 2021-09-10 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Recurrent Wheezes
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
wheezing" is defined as a musical sound caused by the passage of air through narrow respiratory tract airways . Recurrent wheeze is defined as three or more episodes of parentally reported wheeze in the past 12 months of Various risk factors are associated with recurrent wheezing and asthma: small airway caliber; decreased lung function at birth; viral respiratory infections; environmental pollution; pets; early daycare attendance; passive smoking; parental history of asthma or atopy; obesity; and socioeconomic factors.

DETAILED DESCRIPTION:
There has been growing recognition of the critical extra-skeletal roles for vitamin D in recent years with an explosion of interest in vitamin D across health disciplines including lung disease. Recently, vitamin D was found to be low in patients with recurrent wheezes.

Vitamin D, whether produced in the skin upon sun exposure or ingested from various dietary sources, is converted in the liver to 25-hydroxyvitamin D [25(OH)D]. The latter is the major circulating form of vitamin D and is thus used for evaluating the vitamin D status of patients . The flesh of fatty fish (such as salmon, tuna, and mackerel) and fish liver oils are among the best sources of vitamin D and the fortified cereals and milk provide adequate amounts as well.

Studies in animal models and humans have demonstrated an association of low vitamin D concentrations with atopy and respiratory tract conditions. The mechanism that explains this association is still unclear. It has been suggested that this mechanism is due to the effects of vitamin D status on the regulation of the immune system.

The vitamin D receptor is expressed in various cells of the immune system, such as macrophages, monocytes, dendritic cells, and natural killer cells, as well as in B and T lymphocytes. Binding of the active form of vitamin D to its receptor leads to an increase in immunomodulatory activity that maintains the balance between the cellular immune response (Th1) and the humoral response (Th2), in addition to stimulating regulatory T cells.

Hypomagnesaemia (serum Mg level <0.74 mmol.L-1) has been also suggested to be associated with increased incidence of wheeze, airway hyperreactivity, and impairment of lung function. The mechanisms of action of magnesium (Mg) on respiratory airways are multiple and include relaxation of airways smooth muscle, bronchodilatation, anticholinergic effect, and stabilization of the mast cells

ELIGIBILITY:
Inclusion Criteria:

* Any child with three or more episodes of parentally reported wheeze aged from 1 month to less than 6 years admitted at pediatric department of Sohag University Hospital.

Exclusion Criteria:

* patients with chronic lung and congenital heart diseases.
* Patients with body mass index (BMI) below 3rd percentile and those ≥ 85th percentile will be excluded to avoid effect of disturbed nutritional status on vitamin D level and occurrence of wheezing.

Ages: 1 Month to 6 Years | Sex: All
Age Groups: Child
Study Population: The study will include any child with three or more episodes of parentally reported wheeze aged from 1 month to less than 6 years admitted at pediatric department of Sohag University Hospital.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Value of serum vitamin D, calcium and magnesium in infants and preschool recurrent wheezers | One year
  Serum vitamin D, calcium and magnesium venous blood sample (3ml) will be obtained from children with recurrent wheezes aged from 1 month to 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

REFERENCES:
- [Background] Douros K, Everard ML. Time to Say Goodbye to Bronchiolitis, Viral Wheeze, Reactive Airways Disease, Wheeze Bronchitis and All That. Front Pediatr. 2020 May 5;8:218. doi: 10.3389/fped.2020.00218. eCollection 2020. PMID 32432064
- [Background] Ly NP, Gold DR, Weiss ST, Celedon JC. Recurrent wheeze in early childhood and asthma among children at risk for atopy. Pediatrics. 2006 Jun;117(6):e1132-8. doi: 10.1542/peds.2005-2271. PMID 16740815
- [Background] de Sousa RB, Medeiros D, Sarinho E, Rizzo JA, Silva AR, Bianca AC. Risk factors for recurrent wheezing in infants: a case-control study. Rev Saude Publica. 2016;50:15. doi: 10.1590/S1518-8787.2016050005100. Epub 2016 May 3. PMID 27143615
- [Background] Yang HK, Choi J, Kim WK, Lee SY, Park YM, Han MY, Kim HY, Hahm MI, Chae Y, Lee KJ, Kwon HJ, Ahn K, Kim J. The association between hypovitaminosis D and pediatric allergic diseases: A Korean nationwide population-based study. Allergy Asthma Proc. 2016 Jul;37(4):64-9. doi: 10.2500/aap.2016.37.3957. PMID 27401310